CLINICAL TRIAL: NCT06458374
Title: Prevalence and Long Tem Follow Up of ATTR Cardiac Amyloidosis in a Selected Population of Patients Operated on Carpal Tunnel Syndrome
Brief Title: ATTR Cardiac Amyloidosis in a Selected Population
Status: Recruiting | Type: Observational
Sponsor: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 715238
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: ATTR Amyloidosis Wild Type; ATTR Gene Mutation; Carpal Tunnel Syndrome; Cardiac Amyloidosis
MeSH Terms: conditions — Carpal Tunnel Syndrome; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients operated for carpal tunnel syndrome (CTS) at Ålesund Hospital (200 patients) will have a biopsy to diagnose ATTR amyloidosis. Patients with positive biopsy will be examined to decide wether they have cardiac amyloidosis. All patients with positive biopsy will be followed closely for 10 years wit echocardiography an clinically.

DETAILED DESCRIPTION:
Biopsy proven ATTR (v/wt) amyloidosis inpatients operated with CTS will undergo standard guidelines recommended examinations as 99mTcDPD SPECT CT, echocardiography, ECG, Holter, genetic testing (v/wt), and lab testing, and CMRI as indicated. Exclusion of light chain disease will be done.

All patients will be followed at least yearly as indicated by guidelines (ESC), and patients with development of cardiac amyloidosis will get standard treatment in accordance with guidelines and as approved by the Norwegian government. All patients will be followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Male > 50 years
* Female > 60 years
* operated CTS at Ålesund Hospital

Exclusion Criteria:

* not consented
* do not speak Norwegian
* secondary cause of CTS as traumatic or rheumatic
* cannot be followed > 5 years due to other medical conditions
* Cardiac disease at time of operation for CTS

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maximum 200 patients operated at Ålesund Hospital for CTS
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-02-28 (Estimated); Study Completion 2039-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of ATTR in CTS | 2 years
  Biopsy proven ATTR
Cardiac involvement in patients with biopsy proven ATTR | 10 years
  Scintigraphic and echocardiographic cardiac involvement possibly cMRI

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Hole, MD, PhD, Principal Investigator — Helse Møre og Romsdal HF and NTNU
Locations (1):
- Ålesund Hospital, Ålesund, Møre og Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No